CLINICAL TRIAL: NCT04684407
Title: Assessment of C-reactive Protein Levels in Acute Apical Abscess Due to Root Canal Infection
Brief Title: C-reactive Protein Levels in Acute Apical Abscess Due to Root Canal Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSI College of Dental Sciences and Research, Madurai (Other)
Responsible Party: Principal Investigator, Dr.Joyson Joe Asir.J, Post graduate student, CSI College of Dental Sciences and Research, Madurai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CSIDentalCMadurai
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Dentoalveolar Abscess
MeSH Terms: conditions — Periapical Abscess

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide (Active Comparator): calcium hydroxide powder is mixed with normal saline and placed as intra-canal medication
  Interventions: Procedure: ROOT CANAL TREATMENT
- Triple antibiotic paste (Experimental): Triple antibiotic paste (TAP)- combination of metronidazole,ciprofloxacin and minocycline mixed in a ratio of 1:1:1 .
  TAP paste is combined with propylene glycol and placed as intra canal medication.
  Interventions: Procedure: ROOT CANAL TREATMENT

INTERVENTIONS:
Procedure: ROOT CANAL TREATMENT — TWO TYPE OF INTRA CANAL MEDICATION PLACEMENT

SUMMARY:
C-reactive protein levels of patients with acute apical abscess are evaluated before and after root canal treatment

DETAILED DESCRIPTION:
In patients with acute apical abscess C-reactive proteins are evaluated before and after root canal treatment. In this intra-canal medications calcium hydroxide and triple antibiotic paste are compared. PAI score of the corresponding tooth is noted .

ELIGIBILITY:
Inclusion Criteria:

patient with acute apical abscess

Exclusion Criteria:

* Teeth with evidence of previous initiated root canal treatment
* History of myocardial infarction, coronary heart disease
* Patients allergic to local anesthetic
* Patients under steroid medication
* Patients who are immunocompromised

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Post root canal C reactive protein level | 2 weeks
  Pre-operative serum c-reactive protein level was measured to which the post operative c-reactive protein level after 2 weeks of root canal treatment are compared.
  The normal serum c-reactive protein level is 0 - 6.00 mg/L.

SECONDARY OUTCOMES:
pain and swelling assessment | 6 months
  pain and swelling reduction after root canal treatment is assessed. . Pain is evaluated using visual analgue scale (VAS) , regarding swellling reduction patient is asked to evaluate subjectively whether the patient profile has returned to normal after the treatment and they were asked how many days it took for the swelling to resolve completely.

CONTACTS AND LOCATIONS:
Locations (1):
- Csi College of Dental Sciences and Research, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No